CLINICAL TRIAL: NCT04450914
Title: Implementing Shared Decision Making (SDM) For Individualized CV Prevention (SDM4IP)
Acronym: SDM4IP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jennifer L. Ridgeway, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-002772
Record Dates: First submitted 2020-06-22; First posted 2020-06-30 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Risk; Cardiovascular Prevention

STUDY DESIGN:
Intervention Model Description: Mixed method, hybrid implementation-effectiveness (Type III) step-wedge clustered randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Health Systems - First Step (Other): Each health system will consist of clinicians who are affiliated with primary care practices and patients who are eligible for CV primary prevention discussions. In the first step, health systems will be assigned to usual care (passive implementation of CV Prevention Choice).
  Interventions: Behavioral: CV Prevention Choice Tool
- Health Systems - Second Step (Other): Each health system will consist of clinicians who are affiliated with primary care practices and patients who are eligible for CV primary prevention discussions. In the second step, health systems (in an order to be determined by randomization and staggered over time) will move into active implementation.
  Interventions: Behavioral: CV Prevention Choice Tool; Behavioral: Implementation Facilitation Strategies
- Health Systems - Third Step (Other): Each health system will consist of clinicians who are affiliated with primary care practices and patients who are eligible for CV primary prevention discussions.In the third step, all health systems will move to maintenance implementation.
  Interventions: Behavioral: CV Prevention Choice Tool

INTERVENTIONS:
Behavioral: CV Prevention Choice Tool — The CV Prevention Choice SDM tool is a shared decision making intervention. It is embedded in the electronic health record and uses EHR data to estimate and display cardiovascular risk for individual patients and then foster conversations between clinicians and patients about available options for preventive care based on individual risk and preferences.
Behavioral: Implementation Facilitation Strategies — During the active implementation stage, health systems will deploy tailored implementation facilitation and other tailored implementation strategies aimed at increasing adoption and use of shared decision making using CV Prevention Choice.
  Arms: Health Systems - Second Step

SUMMARY:
Cardiovascular (CV) disease is the #1 cause of premature mortality and substantial morbidity in the U.S. Despite clinical guidelines, most clinical interventions are implemented in people at relatively lower CV risk, and few among people at the highest risk. Shared decision making (SDM) can mitigate the risk-treatment paradox by reducing risk blindness and lack of fit of the preventive regimen, but the adoption of SDM in routine clinical care is incomplete. This study addresses SDM adoption of a CV prevention SDM tool in three health systems.

DETAILED DESCRIPTION:
The primary prevention of cardiovascular (CV) events is often more intense in individuals at lower risk and vice versa (the so called "risk-treatment paradox") in part due to unawareness of each person's CV risk, of their preferences for prevention interventions, and of their feasibility in each person's daily life. Clinical practice guidelines recommend that clinicians and patients work together to arrive at an effective and feasible prevention plan that is congruent with each person's CV risk and informed preferences, a process called shared decision making (SDM). Despite the availability of an innovative and effective tool that estimates CV risk, shows the impact and features of available lifestyle and pharmacological preventive interventions, and thus can facilitate CV treatment discussions between clinicians and patients, this type of SDM does not routinely happen in practice.

The challenge therefore is to identify strategies to increase adoption of this type of SDM in real-world clinical practices. This 4-year study - proposed by a multidisciplinary team with expertise in preventive cardiology, SDM, and implementation science - aims to integrate an SDM tool (the CV Prevention Choice tool) in the primary care practices of three diverse health care systems in the U.S. and study both the tool and tailored strategies that foster its adoption and routine use. The study will use a mixed method, hybrid implementation-effectiveness (Type III) step-wedge clustered randomized trial design to determine:

* Implementation effectiveness (Aim 1) by evaluating the settings (including local workflow and policies) in which the CV Prevention Choice tool is implemented and the engagement of users in implementation strategies; implementation outcomes (e.g., reach, adoption) associated with these strategies; and how implementation fosters routine adoption of SDM and the CV Prevention Choice tool in primary care practices, and
* SDM effectiveness (Aim 2) estimated by the extent to which individual CV prevention plans are feasible and congruent with each person's estimated CV risk and preferences.

The investigators hypothesize that efforts to assess local needs and use them to develop tailored implementation approaches will foster greater adoption of SDM in practice. They further hypothesize that individual preventive care plans will be congruent with estimated risk when clinicians adopt the SDM tool. The broad goal is to promote patient-centered care that effectively reduces the substantial burden of CV disease among Americans. By the project's end, the investigators expect to have (a) identified the most effective implementation strategies to embed SDM in routine practice and (b) estimated the effectiveness of SDM to achieve feasible and risk-concordant CV prevention in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Clinician Participants: All clinicians who are affiliated with a participating primary care practice and care for adult patients eligible for CV prevention will be invited to participate.
* Patient Participants: Adult patients (ages 40-75 years) with or without diabetes who have not experienced an atherothrombotic clinical event and receive preventive care at a participating primary care practice will be eligible to participate.

Exclusion Criteria:

- Individuals who do not speak English or have any sort of cognitive deficit that would impact their ability to consent to participate in the study will not be invited to participate.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112127 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Reach metrics | Q1/Year 2 through Q3/Year 4
  Proportion of eligible clinicians who accessed CV Prevention Choice (among all eligible clinicians), as indicated by EHR user metrics. Higher proportions indicate greater reach.
Effectiveness perceptions | Q1/Year 2 through Q3/Year 4
  Qualitative findings of the perceptions of tool effectiveness, as assessed through interviews and focus groups with eligible clinicians.
Adoption metrics | Q1/Year 2 through Q3/Year 4
  Proportion of eligible clinicians that used CV Prevention Choice in encounters identified in the EHR as being eligible for a CV preventive care discussion (among all eligible visits), as indicated by EHR user metrics. Higher proportions indicate greater adoption.
Adoption perceptions | Q1/Year 2 through Q3/Year 4
  Qualitative findings of reasons for adoption of or failure to adopt CV Prevention Choice, as assessed through interviews and focus groups with eligible clinicians.
Implementation fidelity | Q1/Year 4 through Q3/Year 4
  A sample of SDM clinical encounters will be audio-video recorded. Recordings will be reviewed and scored according to a five-point SDM fidelity checklist. Higher scores indicate greater fidelity to the core components of SDM.
Implementation SDM quality | Q1/Year 4 through Q3/Year 4
  Adherence to SDM quality will be assessed among a sample of patients with SDM clinical encounters using the Shared Decision Making Questionnaire (SDM-Q-9) questionnaire. Higher scores are indicative of higher levels of SDM occurring in the encounter. Range of scores is 0 to 100.
Implementation care quality | Q1/Year 4 through Q3/Year 4
  Care quality will be assessed among a sample of patients with SDM clinical encounters using the 10-item CARE Patient Feedback Measure. Higher scores are indicative of higher patient reported relational empathy in the consultation. Range of scores is 10 to 50.
Maintenance metrics | Q1/Year 4 through Q3/Year 4
  Change in CV PREVENTION CHOICE use, as indicated by EHR user metrics for eligible clinicians, at the start and end of the maintenance stage. Equivalent or higher use at the end of the maintenance stage indicates maintenance of the tool as part of routine practice.
Maintenance self-report | Q1/Year 4 through Q3/Year 4
  The NoMAD questionnaire will be administered to clinicians to assess normalization of CV Prevention Choice into practice. The NoMAD questionnaire is a continuous outcome converted to a 0-100 point scale, where higher scores indicate higher levels or normalization of CV Prevention Choice into routine care.

SECONDARY OUTCOMES:
SDM Effectiveness | Q1/Year 2 through Q3/Year 4
  The assessment of statin prescription post encounter of interest is congruent with the patient estimated CV Risk based off EHR data.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ridgeway, PhD, Principal Investigator — Mayo Clinic; Victor Montori, MD, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Wellstar Health System, Marietta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - Altru Health System, Grand Forks, North Dakota
  - VHC Health, Arlington, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ridgeway JL, Branda ME, Gravholt D, Brito JP, Hargraves IG, Hartasanchez SA, Leppin AL, Gomez YL, Mann DM, Nautiyal V, Thomas RJ, Behnken EM, Torres Roldan VD, Shah ND, Khurana CS, Montori VM. Increasing risk-concordant cardiovascular care in diverse health systems: a mixed methods pragmatic stepped wedge cluster randomized implementation trial of shared decision making (SDM4IP). Implement Sci Commun. 2021 Apr 21;2(1):43. doi: 10.1186/s43058-021-00145-6. PMID 33883035